CLINICAL TRIAL: NCT00486811
Title: A Randomized Double-blind, Placebo- and Active-control, Parallel-arm, Phase III Trial With Controlled Adjustment of Dose to Evaluate the Efficacy and Safety of CG5503 Prolonged Release (PR) in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee.
Brief Title: A Study to Evaluate the Efficacy and Safety of CG5503 Prolonged Release (PR) in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 335862; 2006-005783-67 (EudraCT Number)
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Pain; Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Pain Assessment; CG5503 PR; Centrally acting analgesic; Placebo; Oxycodone; Chronic Pain due to knee Osteoarthritis; Tapentadol
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matching Placebo (twice daily) (Placebo Comparator): The starting dose of placebo was matched with the active treatment arms taken twice daily for the first 3 days. The dose was then increased to match the active treatments for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days as in the active treatment arms. Dose decreases were allowed without time restrictions.
  Interventions: Drug: Matching Placebo (twice daily)
- Tapentadol ER (100 to 250 mg twice daily) (Experimental): The starting dose was tapentadol ER 50 mg twice daily for 3 days. The dose was then increased to 100 mg tapentadol ER twice daily for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days. Dose decreases were allowed without time restrictions.
  Interventions: Drug: Tapentadol ER (100 to 250 mg twice daily)
- Oxycodone CR (20 to 50 mg twice daily) (Active Comparator): The starting dose was oxycodone CR 10 mg twice daily for 3 days. The dose was then increased to 20 mg oxycodone CR twice daily for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days. Dose decreases were allowed without time restrictions.
  Interventions: Drug: Oxycodone CR (20 to 50 mg twice daily)

INTERVENTIONS:
Drug: Tapentadol ER (100 to 250 mg twice daily) — 50, 100, 150, 200, 250 mg twice a day (BID) during 15 weeks (3 weeks titration and 12 weeks maintenance)
  Arms: Tapentadol ER (100 to 250 mg twice daily)
Drug: Matching Placebo (twice daily) — Matching Placebo during 15 weeks (3 weeks titration and 12 weeks maintenance)
  Arms: Matching Placebo (twice daily)
Drug: Oxycodone CR (20 to 50 mg twice daily) — 10, 20, 30, 40, 50 mg twice a day (BID) during 15 weeks (3 weeks titration and 12 weeks maintenance)
  Arms: Oxycodone CR (20 to 50 mg twice daily)

SUMMARY:
The purpose of this study is to evaluate whether tapentadol (CG5503) prolonged-release (PR) tablets at doses of 100-250 mg twice daily provide a better pain relief in patients with moderate to severe chronic pain due to osteoarthritis of the knee than a placebo (a medication without active substance). In addition the tolerability of CG5503 PR will be assessed. One third of the patients will receive CG5503 and one third will receive placebo. For further comparison one third of the patients will receive oxycodone controlled release (CR) at doses of 20-50 mg twice daily which is an active approved pain medication. Please note that tapentadol ER (Extended Release) and tapentadol PR (Prolonged Release) are identical and used interchangeably. This is due to United States of America and European naming conventions.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to patients by chance), double-blind (neither patient nor investigator knows which patient gets which study medication, i.e. CG5503, placebo, oxycodone), placebo and active control study. The primary objective is to evaluate the efficacy and safety of orally administered tapentadol (CG5503) prolonged-release (PR) at doses of 100-250 mg (base) twice daily in patients with moderate to severe chronic pain from osteoarthritis (OA) of the knee. The study will consist of five periods: screening (to assess eligibility), washout (3-7 days with determination of a baseline pain intensity), titration (of dose over 3 weeks to the optimal individual level), maintenance (investigational drug intake for 12 weeks with adjustments allowed), and follow-up (2 weeks after end of treatment). The study hypothesis is that the study drug will be more effective than placebo in reducing patients' pain intensity. The secondary objectives include the collection of pharmacokinetic (related to how the body absorbs, distributes, changes and excretes the drug) information for dose verification. The efficacy objectives will be assessed by comparing the baseline pain level to the pain level during the maintenance period. This will be done by looking at the patients' pain diary information (electronic diaries).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with osteoarthritis of the knee based on the American College of Rheumatology (ACR) criteria and functional capacity class of I- III;
* Patients taking analgesic medications for at least 3 months prior to screening and dissatisfied with their current therapy;
* Patients requiring opioid treatment must be taking daily doses of opioid- based analgesic, equivalent to <160 mg of oral morphine;
* Baseline score of >=5 on an 11-point numeric rating scale, calculated as the average pain intensity during the last 3 days prior to randomization.

Exclusion Criteria:

* History of alcohol and/or drug abuse in Investigator's judgment;
* Chronic hepatitis B or C, or HIV, presence of active hepatitis B or C within the past 3 months;
* Life-long history of seizure disorder or epilepsy;
* History of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated;
* Uncontrolled hypertension;
* Patients with severely impaired renal function;
* Patients with moderate to severely impaired hepatic function or with laboratory values reflecting inadequate hepatic function,
* Treatment with neuroleptics, monoamine oxidase inhibitors, serotonin norepinephrine reuptake inhibitors (SNRI), tricyclic antidepressants, anticonvulsants, or anti-parkinsonian drugs, treatment with any other analgesic therapy than investigational medication or rescue medication during the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Serrie, Dr., Principal Investigator — C.E.T.D Hôpital Lariboisière, Paris, France
Locations (100):
- Austria (6):
  - Site 043005, Innsbruck
  - Site 043006, Mitterdorf
  - Site 043002, Salzburg
  - Site 043001, Vienna
  - Site 043004, Vienna
  - Site 043003, Wiener Neustadt
- Croatia (5):
  - Site 385003, Karlovac
  - Site 385001, Osijek
  - Site 385004, Sisak
  - Seite 385005, Zagreb
  - Site 385002, Zagreb
- Germany (10):
  - Site 049002, Berlin
  - Site 049008, Berlin
  - Site 049010, Berlin
  - Site 049003, Dresden
  - Site 049004, Frankfurt
  - Site 049007, Hamburg
  - Site 049001, Leipzig
  - Site 049005, Magdeburg
  - Site 049009, Schwerin
  - Site 049006, Wiesbaden
- Hungary (8):
  - Site 036003, Budapest
  - Site 036005, Budapest
  - Site 036006, Budapest
  - Site 036009, Budapest
  - Site 036008, Debrecen
  - Site 036004, Kecskemét
  - Site 036007, Kecskemét
  - Site 036002, Visegrád
- Italy (4):
  - Site 039002, Chieti
  - Site 039003, Milan
  - Site 039004, Pavia
  - Site 039001, Perugia
- Latvia (3):
  - Site 371002, Bauska
  - Site 371004, Riga
  - Site 371005, Riga
- Netherlands (5):
  - Site 031008, Eindhoven
  - Site 031003, Losser
  - Site 031006, Oude Pekela
  - Site 031004, s'Hertogenbosch
  - Site 031007, Spijkenisse
- Poland (11):
  - Site 048007, Bielsko-Biala
  - Site 048005, Gmina Końskie
  - Site 048006, Katowice
  - Site 048004, Krakow
  - Site 048001, Lublin
  - Site 048008, Mielec
  - Site 048003, Piekary Śląskie
  - Site 048010, Rzeszów
  - Site 048009, Warsaw
  - Site 048002, Wroclaw
  - Site 048011, Wroclaw
- Portugal (7):
  - Site 351001, Coimbra
  - Site 351003, Faro
  - Sites 351008, Funchal
  - Site 351005, Guimarães
  - Site 351004, Lisbon
  - Site 351009, Lisbon
  - Site 351002, Ponta Delgada
- Romania (10):
  - Site 040001, Bucharest
  - Site 040002, Bucharest
  - Site 040005, Bucharest
  - Site 040006, Bucharest
  - Site 040007, Bucharest
  - Site 040008, Bucharest
  - Site 040009, Bucharest
  - Site 040011, Bucharest
  - Site 040004, Campulung Muscel
  - Site 040010, Craiova
- Slovakia (5):
  - Site 421005, Banská Bystrica
  - Site 421001, Košice
  - Site 421003, Poprad
  - Site 421004, Prešov
  - Site 421002, Rimavská Sobota
- Spain (12):
  - Site 034002, Alicante
  - Site 034009, Benidorm
  - Site 034005, L'Hospitalet de Llobregat
  - Site 034007, La Roca del Vallès
  - Site 034015, Málaga
  - Site 034008, Móstoles
  - Site 034003, Oviedo
  - Site 034013, Oviedo
  - Site 034016, Seville
  - Site 034001, Torrelavega
  - Site 034012, Valencia
  - Site 034004, Vic
- United Kingdom (14):
  - Site 044012, Birmingham
  - Site 044004, Blackpool
  - Site 044009, Bradford
  - Site 044013, Cardiff
  - Site 044002, Chesterfield
  - Site 044018, Chorley
  - Site 044005, Ecclesfield
  - Site 044008, Falkirk
  - Site 044001, Kenton
  - Site 044006, London
  - Site 044011, London
  - Site 044016, Reading
  - Site 044003, Solihull
  - Site 044007, Woolpit

REFERENCES:
- [Derived] Etropolski M, Kuperwasser B, Flugel M, Haufel T, Lange B, Rauschkolb C, Laschewski F. Safety and tolerability of tapentadol extended release in moderate to severe chronic osteoarthritis or low back pain management: pooled analysis of randomized controlled trials. Adv Ther. 2014 Jun;31(6):604-20. doi: 10.1007/s12325-014-0128-6. Epub 2014 Jul 2. PMID 24985410
- [Derived] Biondi DM, Xiang J, Etropolski M, Moskovitz B. Evaluation of blood pressure and heart rate in patients with hypertension who received tapentadol extended release for chronic pain: a post hoc, pooled data analysis. Clin Drug Investig. 2014 Aug;34(8):565-76. doi: 10.1007/s40261-014-0209-y. PMID 24916058
- [Derived] Etropolski M, Lange B, Goldberg J, Steup A, Rauschkolb C. A pooled analysis of patient-specific factors and efficacy and tolerability of tapentadol extended release treatment for moderate to severe chronic pain. J Opioid Manag. 2013 Sep-Oct;9(5):343-56. doi: 10.5055/jom.2013.0177. PMID 24353047
- [Derived] Merchant S, Provenzano D, Mody S, Ho KF, Etropolski M. Composite measure to assess efficacy/gastrointestinal tolerability of tapentadol ER versus oxycodone CR for chronic pain: pooled analysis of randomized studies. J Opioid Manag. 2013 Jan-Feb;9(1):51-61. doi: 10.5055/jom.2013.0147. PMID 23709304
- [Derived] Afilalo M, Morlion B. Efficacy of tapentadol ER for managing moderate to severe chronic pain. Pain Physician. 2013 Jan;16(1):27-40. PMID 23340531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on 04 June 2007 and the last participant out was on 18 July 2008.
Groups:
- Placebo Matching: Drug: Matching Placebo (twice daily)
  The starting dose of placebo was matched with the active treatment arms taken twice daily for the first 3 days. The dose was then increased to match the active treatments for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days as in the active treatment arms. Dose decreases were allowed without time restrictions.
- Tapentadol ER: Tapentadol ER (100 to 250 mg twice daily) The starting dose was tapentadol ER 50 mg twice daily for 3 days. The dose was then increased to 100 mg tapentadol ER twice daily for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days. Dose decreases were allowed without time restrictions.
  Tapentadol ER 50, 100, 150, 200 or 250 mg twice a day (BID) during 15 weeks were dosed by participants (3 weeks titration and 12 weeks maintenance).
- Oxycodone CR: Oxycodone CR (20 to 50 mg twice daily).
  The starting dose was oxycodone CR 10 mg twice daily for 3 days. The dose was then increased to 20 mg oxycodone CR twice daily for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days. Dose decreases were allowed without time restrictions. Oxycodone doses were thus 10, 20, 30, 40 or 50 mg twice a day (BID) during 15 weeks were dosed by participants (3 weeks titration and 12 weeks maintenance).
Period: Overall Study
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Started | 337 | 320 (One participant was not eligible to be dosed.) | 333 (Two participants were not eligible to be dosed.)
Completed | 215 | 179 | 119
Not Completed | 122 | 141 | 214
Not completed — Adverse Event | 28 | 60 | 135
Not completed — Lack of Efficacy | 34 | 14 | 7
Not completed — Lost to Follow-up | 4 | 6 | 4
Not completed — Withdrawal by Subject | 33 | 44 | 58
Not completed — Study drug non-compliant | 5 | 6 | 3
Not completed — All other | 18 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Oxycodone CR: Oxycodone CR (20 to 50 mg twice daily).
  The starting dose was oxycodone CR 10 mg twice daily for 3 days. The dose was then increased to 20 mg oxycodone CR twice daily for at least 4 days. Thereafter, during the titration and maintenance phase participants were allowed to increase the dose every 3 days. Dose decreases were allowed without time restrictions. Oxycodone doses were thus 10, 20, 30, 40 or 50 mg twice a day (BID) were dosed by participants during 15 weeks (3 weeks titration and 12 weeks maintenance).
- Total: Total of all reporting groups
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR | Total
Number analyzed (Participants) | 337 | 319 | 331 | 987
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.35) | 62.4 (9.35) | 61.8 (9.09) | 62.1 (9.26)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 194 | 194 | 211 | 599
  >=65 years | 143 | 125 | 120 | 388
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 231 | 219 | 707
  Male | 80 | 88 | 112 | 280
Region of Enrollment [Number; unit: participants]
  Portugal | 8 | 4 | 3 | 15
  Slovakia | 7 | 8 | 9 | 24
  Spain | 29 | 23 | 25 | 77
  Austria | 14 | 12 | 15 | 41
  United Kingdom | 23 | 24 | 28 | 75
  Hungary | 36 | 35 | 34 | 105
  Poland | 11 | 11 | 13 | 35
  Romania | 107 | 103 | 104 | 314
  Croatia | 12 | 9 | 8 | 29
  Germany | 58 | 60 | 59 | 177
  Latvia | 24 | 21 | 24 | 69
  Netherlands | 8 | 9 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Average Pain Intensity Overall in the 12-week Maintenance Period of the Daily Pain Intensity on an 11-point Numeric Rating Scale (NRS).
Description: For this twice daily pain assessment, the participants were required to indicate the level of pain experienced over the previous 12 hours on an 11-point Numeric Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The lower the value the less pain in the treatment group. Negative values indicate a reduction in pain.
Time Frame: Change from baseline over the 12 week Maintenance Period
Population: Intent-to-treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 337 | 319 | 331
Units on a scale | -2.2 (2.06) | -2.5 (2.18) | -2.1 (2.17)

2. Secondary Outcome: Change From Baseline of the Average Pain Intensity Based on an 11-point Numerical Rating Scale (NRS) Over the Last Week of the Maintenance Period at Week 12.
Description: The twice daily pain assessments were averaged. The participants were to indicate their pain on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The lower the value the less pain intensity.
Time Frame: Change from Baseline to Week 12 of the Maintenance Period
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 336 | 319 | 331
Units on a scale | -2.5 (2.30) | -2.7 (2.4) | -2.3 (2.36)

3. Secondary Outcome: Patient Global Impression of Change
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of 12 week maintenance period
Population: Intention to treat (ITT). Last observation carried forward (LOCF). Assessments obtained more than one day after end of treatment were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 294 | 248 | 212
participants
  Very Much Improved | 33 | 40 | 25
  Much Improved | 94 | 99 | 65
  Minimally Improved | 76 | 61 | 51
  No Change | 59 | 22 | 30
  Minimally Worse | 15 | 9 | 19
  Much Worse | 14 | 14 | 19
  Very Much Worse | 3 | 3 | 3

4. Secondary Outcome: Change From Baseline in the Western Ontario McMaster Questionnaire (WOMAC) Global Score Assessing Pain, Disability and Joint Stiffness of the Knee Over the Last Week of the Maintenance Period at Week 12
Description: Change from baseline to week 12 of Western Ontario McMaster Questionnaire (WOMAC) Global Score: WOMAC is measured with a Likert ordinal scale (the participant gives one of 5 possible answers) from 0 to 4. Higher scores indicate that a symptom is bothersome and physically disabling.
Time Frame: Change from baseline to week 12 of the maintenance period
Population: Intention to treat (ITT). No imputation performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 218 | 183 | 114
units on a scale | -1.0 (0.92) | -1.0 (0.90) | -1.1 (0.83)

5. Secondary Outcome: Time to Treatment Discontinuation Due to Lack of Efficacy
Description: The median time to treatment discontinuation due to lack of efficacy from baseline to endpoint.
Time Frame: Baseline to week 12 of the maintenance period
Population: Intention to treat (ITT) The results for median and interquartile ranges were not estimated as an insufficient number of participants discontinued due to lack of efficacy to estimate values.
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in the Health Survey Scores Form (SF-36)
Description: The Scores Form 36 (SF-36) includes several brief board questions on 8 aspects, (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. A higher score indicates an improvement in health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state.
Time Frame: Change From Baseline to Week 12 of the Maintenance Period
Population: The number indicate the available responses. For certain categories, e.g. Physical Functioning only 318 participants in the tapentadol treatment were analyzed and in the General Health analysis only 328 oxycodone- and 336 placebo-treated participants were available. Intention to treat (ITT). Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 337 | 319 | 331
units on a scale
  Physical Functioning | 11.1 (23.00) [0 to 0] | 11.70 (22.91) [-1.82 to 4.25] | 9.5 (18.65) [-4.18 to 1.84]
  Role-Physical | 18.7 (45.63) [0 to 0] | 20.8 (43.32) [-5.64 to 5.48] | 13.8 (40.96) [-11.12 to -0.08]
  Bodily Pain | 15.4 (22.01) [0 to 0] | 19.1 (20.92) [-0.29 to 5.75] | 13.9 (20.41) [-5.04 to 0.95]
  General Health | 6.8 (17.07) [0 to 0] | 6.8 (17.56) | 4.8 (15.05)
  Vitality | 6.8 (21.37) [0 to 0] | 7.1 (19.40) | 3.8 (18.40)
  Social Functioning | 7.5 (25.76) [0 to 0] | 9.2 (24.30) | 4.9 (22.91)
  Role-Emotional | 7.9 (48.63) [0 to 0] | 11.1 (45.74) | 5.0 (38.95)
  Mental Health | 6.3 (19.39) [0 to 0] | 3.7 (18.02) | 2.7 (16.98)

7. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome Over Time
Description: The participant scored the EuroQol-5. This is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. The positive values indicate that during the study the health status improved.
Time Frame: Comparison of Baseline to Week 12 of the Maintenance Period
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: Index value
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 337 | 319 | 331
Index value | 0.2 (0.02) | 0.2 (0.02) | 0.1 (0.01)

8. Secondary Outcome: Sleep Questionnaire: Change From Baseline in Sleep Latency Time in Hours to the Last Week of the Maintenance Period.
Description: The Sleep Questionnaire addressed the following question: "How long after bedtime/lights out did you fall asleep last night(hours)?". The mean change from baseline to 12 weeks was studied. Decrease in time, measured in hours, indicates an improvement.
Time Frame: Week 12 of the maintenance period compared to baseline
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 327 | 305 | 314
hours | 0.4 (3.68) | 0.2 (2.33) | 0.2 (2.14)

9. Secondary Outcome: Sleep Questionnaire: Amount of Time Slept in Hours
Description: The Sleep Questionnaire addressed the following question: "How long did you sleep last night?". The mean change for the number of hours slept during the night before from baseline to 12 weeks was studied.
Time Frame: Baseline to Week 12 of the maintenance period
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 327 | 305 | 314
hours | 0.2 (2.10) | 0.2 (2.29) | 0.3 (2.01)

10. Secondary Outcome: Sleep Questionnaire: Number of Awakenings During Sleep
Description: The Sleep Questionnaire addressed the following question: "How many times did you wake up during the night?". Sleep was assessed by the subject once a week during the entire double-blind treatment period. Reported are the baseline and end of maintenance period. Generally the less the number of awakenings the better the sleep.
Time Frame: Week 12 of the maintenance period compared with baseline
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF). The number reflects the number of participants that had the specified awakenings.
Measure: Number; unit: participants
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 337 | 319 | 328
participants
  No awakening during night baseline | 32 | 33 | 29
  No awakening during night end point | 55 | 44 | 46
  1 awakening per night baseline | 56 | 53 | 57
  1 awakening per night end point | 89 | 92 | 67
  2 awakening per night baseline | 102 | 88 | 85
  2 awakening per night end point | 84 | 94 | 89
  3 awakening per night baseline | 82 | 66 | 77
  3 awakening per night end point | 66 | 46 | 61
  4 awakening per night baseline | 33 | 39 | 38
  4 awakening per night end point | 21 | 22 | 42
  5 or more awakenings per night baseline | 22 | 26 | 28
  5 or more awakenings per night end point | 22 | 21 | 23

11. Secondary Outcome: Number of Participants Reporting a Category From the Quality of Sleep (Sleep Questionnaire)
Description: The Sleep Questionnaire addressed the following question: "Please rate the overall quality of your sleep last night?" The quality of sleep at baseline and prior to completion of treatment are reported. The participant can choose one of the following options: Excellent, good, fair and poor.
Time Frame: Week 12 of the maintenance period compared to baseline
Population: Intention to treat (ITT). Last Observation Carried Forward (LOCF). The number of participants reporting the appropriate sleep quality category are shown.
Measure: Number; unit: participants
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 337 | 319 | 328
participants
  Excellent at baseline | 11 | 8 | 5
  Excellent at end point | 10 | 15 | 19
  Good at baseline | 134 | 122 | 118
  Good at end point | 174 | 177 | 158
  Fair at baseline | 146 | 138 | 151
  Fair at end point | 124 | 107 | 125
  Poor at baseline | 36 | 37 | 40
  Poor at end point | 29 | 20 | 26

12. Secondary Outcome: Patient Assessment of Constipation Symptoms (PAC-SYM) Over Time
Description: The Constipation Assessment (PAC-SYM) is a 12-item self-report questionnaire that assesses the severity of symptoms of constipation. Participants are asked "How severe have each of these symptoms been in the last two weeks?" e.g. "Pain in your stomach". There are 3 subscales: 4 questions on Abdominal symptoms, 3 on rectal symptoms and 5 on stool symptoms. Responses are rated on a 5-point Likert scale ranging from 0 (absence of symptom) to 4 (very severe symptoms). If the changes in the overall or subscale scores are positive then there is a worsening in symptoms associated with constipation.
Time Frame: Change from Baseline to Week 12 of the Maintenance Period
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 285 | 235 | 197
Units on a scale
  Overall abdominal subscale change | -0.1 (0.69) | 0.1 (0.78) | 0.3 (0.85)
  Overall rectal subscale change | 0.0 (0.52) | 0.1 (0.65) | 0.4 (0.81)
  Overall stool subscale change | 0.0 (0.74) | 0.2 (0.83) | 0.6 (0.97)
  Overall PAC-SYM score change | 0.0 (0.56) | 0.1 (0.64) | 0.4 (0.72)

ADVERSE EVENTS:
Time Frame: Baseline to week 12 of the maintenance period
Arm/Group | Placebo Matching | Tapentadol ER | Oxycodone CR
Serious Adverse Events (participants affected / at risk) | 4/337 | 2/319 | 13/331
Other Adverse Events (participants affected / at risk) | 187/337 | 214/319 | 281/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching (N=337) | Tapentadol ER (N=319) | Oxycodone CR (N=331)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 3
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0
Tachycardia Paroxysmal (Cardiac disorders) | 0 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 0 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine Leimyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching (N=337) | Tapentadol ER (N=319) | Oxycodone CR (N=331)
Nausea (Gastrointestinal disorders) | 21 | 65 | 123
Constipation (Gastrointestinal disorders) | 31 | 56 | 114
Vomiting (Gastrointestinal disorders) | 13 | 32 | 86
Dry Mouth (Gastrointestinal disorders) | 7 | 19 | 13
Diarrhoea (Gastrointestinal disorders) | 15 | 14 | 26
Abdominal Pain Upper (Gastrointestinal disorders) | 20 | 11 | 15
Addominal Pain (Gastrointestinal disorders) | 7 | 4 | 18
Dizziness (Nervous system disorders) | 29 | 70 | 88
Somnolence (Nervous system disorders) | 13 | 34 | 48
Headache (Nervous system disorders) | 31 | 33 | 27
Fatigue (General disorders) | 11 | 25 | 33
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 29 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4 | 36
Vertigo (Ear and labyrinth disorders) | 7 | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor and the Sponsor's designee reserves the right to review any publication pertaining to the trial at least 30 days before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.